CLINICAL TRIAL: NCT02580721
Title: The Influence of Mucosal Tissue Thickness on Soft and Hard Tissue Changes Around Implants. A Randomized Controlled Clinical Study
Brief Title: The Influence of Mucosal Tissue Thickness on Soft and Hard Tissue Changes Around Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, M.Emre Benlidayi, Associate Professor, Cukurova University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: I-BI-15-003
Record Dates: First submitted 2015-10-11; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Post-osseointegration Biological Failure of Dental Implant; Alveolar Bone Loss
Keywords: mucosal tissue thickness; dental implant; marginal bone loss; soft tissue
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Thick mucosal tissue (Active Comparator): Implants with platform switching (Astra Tech Implant System EV) will be placed and cover screws will be inserted.
  Interventions: Device: Dentsply Astra Tech Implant System EV
- Thin mucosal tissue (Experimental): Implants with platform switching (Astra Tech Implant System EV) will be placed and cover screws will be inserted.
  Interventions: Device: Dentsply Astra Tech Implant System EV
- Thickened mucosa with connective tissue (Experimental): Implants with platform switching (Astra Tech Implant System EV) will be placed and cover screws will be inserted. Soft tissue augmentation will be performed with sub epithelial connective tissue graft.
  Interventions: Device: Dentsply Astra Tech Implant System EV
- Thickened mucosa with ADM (Experimental): Implants with platform switching (Astra Tech Implant System EV) will be placed and cover screws will be inserted. Acellular dermal matrix, thick 1 x 4 cm will be used for vertical soft tissue augmentation.
  Interventions: Device: Dentsply Astra Tech Implant System EV

INTERVENTIONS:
Device: Dentsply Astra Tech Implant System EV — Dentsply Astra Tech Implant System EV will be placed

SUMMARY:
Crestal bone and soft tissue stability around implants is an important issue in implant dentistry. Initial vertical mucosal tissue thickness was shown to be one of the factors having impact on bone stability. However, there is lack of data in the literature regarding the relationship between mucosal thickness and marginal bone loss around implants. Berglundh and Lindhe in an animal study reported that thin mucosal tissue causes significantly more crestal bone resorption around implants. In addition, clinical research regarding the effects of tissue thickness on bone and soft tissue stability around implants is lacking. The aim of this clinical study is to evaluate the influence of mucosal tissue thickness on soft and hard tissue changes around implants.

DETAILED DESCRIPTION:
The objectives of this clinical study are;

* to evaluate the influence of mucosal tissue thickness on periimplant soft and hard tissue changes.
* to evaluate whether acellular dermal matrix (ADM) derived allogenic membrane or subepithelial connective tissue grafts performed at implant placement could be effective in vertical soft tissue augmentation.
* to evaluate the influence of vertical soft tissue augmentation with acellular dermal matrix or subepithelial connective tissue grafts on soft and hard tissue changes around implants with platform switching after 1 year of loading.

Partially edentulous patients in the posterior lower jaw area requiring implant treatment will be recruited for this study. There will be four groups in the study with 35 patients in each group.

Inclusion criteria will be; (1) >18 years of age; (2) no medical contraindication for implant surgery; (3) missing teeth in the posterior mandibular area requiring two implants supported three unit bridge prosthetic restoration; (4) fully healed bone sites (at least 3 months after extraction) (5) minimum of 6mm bone width and 10 mm bone height above inferior alveolar canal; (6) healthy soft tissue; (7) minimum 2mm keratinized gingiva; (8) no bone augmentation procedures before and during implant placement. The patients will be excluded if they will not meet inclusion criteria and additionally have (1) poor oral hygiene; (2) uncontrolled periodontitis (3) smoking Ethical approval was taken from Cukurova University Ethical Committee and the patients will sign informed consent form before participating in the study. Cone beam computerized tomography will be taken from all patients in order to evaluate the future implant sites. Patients will be enrolled if they fulfill the inclusion criteria. Patients will be excluded if they will not meet inclusion criteria and additionally have exclusion criteria. Two implants per patient will be placed. The prosthetic restorations will be performed as three unit bridge with two supported implants. These two implants in the premolar and molar regions will be included into the study and evaluated independently.

One hour prior to surgery the patients will receive prophylactic dose of 1 g amoxicillin+clavulanic acid. All surgical procedures will be performed by two experienced surgeons under local anesthesia. A mid-crestal incision on the center of edentulous ridge will be performed, leaving at least width of 2 mm keratinized tissues buccally. Next, a full-thickness buccal flap will be raised, while lingual part will not be elevated to ensure direct visibility. Vertical thickness of soft tissues will be measured with 1.0 mm marked periodontal probe. The probe will be positioned in an upright position to the bone crest in the center of the future implant placement. After measurement, lingual flap will be raised to completely expose the implantation site. If vertical soft tissue thickness is 2 mm or less, tissues will be considered as thin. If soft tissue thickness is more than 2mm, tissues will be considered as thick. There will be four groups in the study.

Group 1: implants placed in naturally thick tissues (>2mm) (control group). Group 2: implants placed in thin tissues (≤2mm) Group 3: vertical soft tissue augmentation in thin tissues (≤2mm) with subepithelial connective tissue graft (SCTG) simultaneously with implant placement.

Group 4: vertical soft tissue augmentation in thin tissues (≤2mm) with AlloDerm® Regenerative Tissue Matrix simultaneously with implant placement.

Implants with platform switching (Astra Tech Implant System EV) will be placed and cover screws will be inserted. In group 3, vertical soft tissue augmentation will be performed with SCTG. In group 4, AlloDerm® RTM, Thick 1 x 4 cm will be used according to manufacturer's recommendations for vertical soft tissue augmentation. The flaps will be closed primarily with 4/0 sutures in all groups.

Patients will be instructed to rinse the operated site with antiseptic mouthwash twice a day and prescribed 1 g of amoxicillin+clavulanic acid twice a day for a week. For pain control, patients will receive 500 mg of flurbiprofen as needed. The sutures will be removed 7-10 days after surgery.

After 3 months of healing second stage surgery will be scheduled under local anesthesia. A mid-crestal incision will be performed in the center of the bone crest. A full-thickness buccal flap will be raised, and thickness of augmented soft tissues over the center of the implant will be measured with a periodontal probe. After raising the lingual flap Astra Tech healing uni EV will be connected to the implant. Flap will be closed with sutures and the sutures will be removed 7 days after surgery. After 14 days of healing Astra Tech uni abutment EV will be connected to the implant and abjutment disconnection will not be performed in order to avoid disruption of the peri-implant seal during abutment unscrewing. Screw retained fixed prosthesis with metal ceramic restoration will be connected to the implant after 6 weeks of healing. Plaque Index (PI), Gingival Index (GI), Probing Pocket Depth (PPD), Bleeding on Probing (BOP), will be evaluated at prosthetic delivery, 6 months and 12 months after loading.

Radiological evaluation and measurements will be performed to calculate the mesial and distal crestal bone changes around implants. Intraoral digital radiographs by using paralleling technique will be taken from patients (i) after implant placement, (ii) after 3 months of healing, (iii) after prosthetic delivery, (iv) after 6 and (v) 12 months of loading. The measurements will be performed using Image J analysis software program (Image J version 1.44-National Institutes of Health, NIH) by an examiner who is unaware of the group assignment. The intra-examiner agreement will be determined by second and third measurements with 1- month interval. The mean difference between measurements will be calculated and the mean of three measurements will be used.

A total of 280 implants in 140 patients with 35 patients in each group will be included in the study according to the results of power analysis. Finally, it will be a patient based study design. Data will be analyzed using SPSS 21.0 (Chicago, IL, USA). Descriptive statistics will be calculated for the measurements as means, SEs, SDs, medians, and range of the measurements. The normality of the distribution will be tested using Kolmogorov Smirnov (P=0.05). One-way ANOVA followed by Tukey HSD tests will be used to compare the group means. As an alternative, Kruskal Wallis H test followed by Mann Whitney U test will be used in case if nonparametric analysis is needed.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. no medical contraindication for implant surgery
3. missing teeth in the posterior mandibular area requiring two implants supported three unit bridge prosthetic restoration
4. fully healed bone sites (at least 3 months after extraction)
5. minimum of 6mm bone width and 10 mm bone height above inferior alveolar canal
6. healthy soft tissue
7. minimum 2mm keratinized gingiva
8. no bone augmentation procedures before and during implant placement.

Exclusion Criteria:

* The patients will be excluded if they will not meet inclusion criteria and additionally have

  1. poor oral hygiene
  2. uncontrolled periodontitis
  3. smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss around implant | The mean change in marginal bone loss from baseline marginal bone level at implant placement to 12 months of implant loading.
  The measurements will be performed using Image J analysis software program (Image J version 1.44-National Institutes of Health, NIH) by an examiner who is unaware of the group assignment. The intra-examiner and inter-examiner agreement will be determined.

SECONDARY OUTCOMES:
Soft tissue changes around implant | Periodontal indexes will be evaluated at 18 weeks after implant placement at prosthetic delivery.
  The measurements will be performed clinically by an examiner who is unaware of the group assignment.
Soft tissue changes around implant | Periodontal indexes will be evaluated at 6 months after implant loading
  The measurements will be performed clinically by an examiner who is unaware of the group assignment.
Soft tissue changes around implant | Periodontal indexes will be evaluated at 12 months after implant loading.
  The measurements will be performed clinically by an examiner who is unaware of the group assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet E Benlidayi, DDS, PhD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University Faculty of Dentistry, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. Influence of thin mucosal tissues on crestal bone stability around implants with platform switching: a 1-year pilot study. J Oral Maxillofac Surg. 2010 Sep;68(9):2272-7. doi: 10.1016/j.joms.2009.08.018. PMID 20605308
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. Reaction of crestal bone around implants depending on mucosal tissue thickness. A 1-year prospective clinical study. Stomatologija. 2009;11(3):83-91. PMID 19996674
- [Background] Berglundh T, Lindhe J. Dimension of the periimplant mucosa. Biological width revisited. J Clin Periodontol. 1996 Oct;23(10):971-3. doi: 10.1111/j.1600-051x.1996.tb00520.x. PMID 8915028
- [Background] Puisys A, Vindasiute E, Linkevciene L, Linkevicius T. The use of acellular dermal matrix membrane for vertical soft tissue augmentation during submerged implant placement: a case series. Clin Oral Implants Res. 2015 Apr;26(4):465-470. doi: 10.1111/clr.12401. Epub 2014 Apr 30. PMID 24779749
- [Background] Bengazi F, Lang NP, Caroprese M, Urbizo Velez J, Favero V, Botticelli D. Dimensional changes in soft tissues around dental implants following free gingival grafting: an experimental study in dogs. Clin Oral Implants Res. 2015 Feb;26(2):176-82. doi: 10.1111/clr.12280. Epub 2013 Oct 24. PMID 24151824
- [Background] Puisys A, Linkevicius T. The influence of mucosal tissue thickening on crestal bone stability around bone-level implants. A prospective controlled clinical trial. Clin Oral Implants Res. 2015 Feb;26(2):123-9. doi: 10.1111/clr.12301. Epub 2013 Dec 9. PMID 24313250
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. The influence of soft tissue thickness on crestal bone changes around implants: a 1-year prospective controlled clinical trial. Int J Oral Maxillofac Implants. 2009 Jul-Aug;24(4):712-9. PMID 19885413